CLINICAL TRIAL: NCT02781324
Title: Use of Ultrasonic Bone Scalpel in Adolescent Idiopathic Scoliosis - Randomized Clinical Trial
Brief Title: Use of Ultrasonic Bone Scalpel in Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-0036
Record Dates: First submitted 2016-05-13; First posted 2016-05-24 (Estimated); Results first posted 2019-06-07 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-12

CONDITIONS: Adolescent Idiopathic Scoliosis; Posterior Spinal Fusion
Keywords: Ultrasonic Bone Scalpel; Adolescent Idiopathic Scoliosis; Posterior Spinal Fusion; Estimated Blood Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasonic Bone Scalpel Group (Experimental): Surgeons will use the ultrasonic bone scalpel, to their discretion, along with standard of care manual devices when performing the posterior spinal fusion.
  Interventions: Procedure: Posterior Spinal Fusion; Device: Ultrasonic Bone Scalpel
- Standard of Care Group (Active Comparator): Surgeons will use, to their discretion, only standard of care manual devices when performing the posterior spinal fusion.
  Interventions: Procedure: Posterior Spinal Fusion

INTERVENTIONS:
Procedure: Posterior Spinal Fusion
Device: Ultrasonic Bone Scalpel
  Arms: Ultrasonic Bone Scalpel Group

SUMMARY:
The primary purpose of this randomized trial is to compare the efficacy of an ultrasonic bone scalpel (or osteotome device) with standard of care surgical instruments during posterior spine fusion with instrumentation.

ELIGIBILITY:
Inclusion Criteria:

1. 10-18 years of age
2. Diagnosis of Adolescent Idiopathic Scoliosis (AIS)
3. Scheduled for a posterior spinal fusion (without Schwab Grade II or higher osteotomy)

Exclusion Criteria:

1. Plan for a posterior column osteotomy of Schwab Grade II or higher
2. Prior spinal surgery
3. Magnetic Resonance Imaging (MRI) abnormalities (such as syrinx and/or chiari malformations)
4. Subjects with medical comorbidities (e.g. heart, lung, kidney disease)
5. Subjects with bleeding diatheses
6. Non-idiopathic etiology for scoliosis

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumeet Garg, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ultrasonic Bone Scalpel Group: Surgeons will use the ultrasonic bone scalpel, to their discretion, along with standard of care manual devices when performing the posterior spinal fusion.
  Posterior Spinal Fusion
  Ultrasonic Bone Scalpel
- Standard of Care Group: Surgeons will use, to their discretion, only standard of care manual devices when performing the posterior spinal fusion.
  Posterior Spinal Fusion
Period: Overall Study
Arm/Group | Ultrasonic Bone Scalpel Group | Standard of Care Group
Started | 33 | 33
Completed | 31 | 31
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasonic Bone Scalpel Group | Standard of Care Group | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31 | 31 | 62
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 30 | 52
  Male | 9 | 1 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21 | 26 | 47
  Hispanic | 5 | 1 | 6
  Black | 1 | 1 | 2
  Asian | 2 | 2 | 4
  Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Estimated Blood Loss/Level
Description: Estimated blood loss is being obtained from the report generated by the cell saver.
Time Frame: Intraoperative
Population: The above 65 patients were analyzed as part of a treated cohort and an intention-to-treat cohort. The discrepancy between the 65 patients with data evaluated and the 66 patients initially consented is explained by 1 patient who withdrew consent from the study. The study team therefore did not feel it was ethical to collect this patient's data.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Ultrasonic Bone Scalpel Group | Standard of Care Group
Number analyzed (Participants) | 32 | 33
mL | 35.21 (18.09) | 38.68 (15.34)

2. Secondary Outcome: Number of Patients With Intraoperative and Postoperative Blood Transfusions in the Ultrasonic Bone Scalpel Group and Standard of Care Group
Description: This outcome measure measures the number of patients with intraoperative and postoperative blood transfusions placed in the Ultrasonic Bone Scalpel Group and the Standard of Care Group.
Time Frame: Intraoperative, Short Term Postoperative (end of procedure until hospital discharge, up to 7 days after surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasonic Bone Scalpel Group | Standard of Care Group
Number analyzed (Participants) | 32 | 33
Participants | 32 | 33

3. Secondary Outcome: Procedure Time (Minutes)
Time Frame: Intraoperative (for duration of the procedure)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ultrasonic Bone Scalpel Group | Standard of Care Group
Number analyzed (Participants) | 32 | 33
minutes | 157.5 (39.46) | 159.7 (36.25)

4. Other Pre Specified Outcome: Preoperative Major Cobb Angle (Degrees)
Description: measured from preoperative radiographs
Time Frame: Preoperative (up to 1 month before scheduled date of surgery)
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Ultrasonic Bone Scalpel Group | Standard of Care Group
Number analyzed (Participants) | 32 | 33
degrees | 49.78 (8.37) | 51.15 (7.7)

5. Other Pre Specified Outcome: Postoperative Major Cobb Angle (Degrees)
Description: Cobb angle is a measurement of the degree of side-to-side spinal curvature used to define Scoliosis. A Cobb angle of 10 degrees is the minimum angle to define scoliosis. Angles of 40-50 degrees or more may require corrective surgery. Cobb angle will be measured from postoperative radiographs
Time Frame: Short Term Postoperative (3 month), Long Term Postoperative (1 year)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Number of Vertebral Levels Fused
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: vertebral levels
Arm/Group | Ultrasonic Bone Scalpel Group | Standard of Care Group
Number analyzed (Participants) | 32 | 33
vertebral levels | 10.53 (2.74) | 10.55 (1.82)

7. Other Pre Specified Outcome: BMI Percentile at Surgery
Time Frame: Preoperative (on day of surgery)
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Ultrasonic Bone Scalpel Group | Standard of Care Group
Number analyzed (Participants) | 32 | 33
percentile | 53.92 (28.42) | 55.7 (25.63)

8. Other Pre Specified Outcome: Weight (kg) at Surgery
Time Frame: Preoperative (on day of surgery)
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Ultrasonic Bone Scalpel Group | Standard of Care Group
Number analyzed (Participants) | 32 | 33
kilograms | 52.45 (10.37) | 54.14 (8.96)

9. Other Pre Specified Outcome: Percent of Participants With Lenke 1 Curve Pattern
Description: Lenke Type 1 is a main thoracic curve pattern, and is the most common pattern observed in cases of adolescent idiopathic scoliosis (AIS). The Lenke Classification System provides surgeons with a simple, accurate, and reproducible way to communicate about scoliosis. It relies on measurements taken from standard x-rays. The surgeon evaluates the x-ray from the front, side, and in bending positions. Each scoliosis curve is then classified in three ways: by the curve type based on the three regions of the spine, a lumbar spine modifier, and a sagittal thoracic modifier. The classification system combines the curve type (1-6) with the lumbar modifier (A, B, C) and the sagittal thoracic modifier (-. N, +) to form the complete classification.
Time Frame: Preoperative (up to 1 month before scheduled date of surgery)
Measure: Number; unit: percentage of participants
Arm/Group | Ultrasonic Bone Scalpel Group | Standard of Care Group
Number analyzed (Participants) | 32 | 33
percentage of participants | 53 | 64

10. Other Pre Specified Outcome: Preoperative Hematocrit
Time Frame: Preoperative (prior to first incision)
Population: one less standard of care participant analyzed because labs were not drawn in designated window.
Measure: Mean (Standard Deviation); unit: grams/deciliter
Arm/Group | Ultrasonic Bone Scalpel Group | Standard of Care Group
Number analyzed (Participants) | 32 | 32
grams/deciliter | 38.24 (5.77) | 36.5 (12.73)

11. Other Pre Specified Outcome: Postoperative Hematocrit
Time Frame: Short Term Postoperative (12-18 hours after procedure)
Population: deviation in numbers due to some postop labs not being drawn and therefore no postop hematocrit values were collected
Measure: Mean (Standard Deviation); unit: grams/deciliter
Arm/Group | Ultrasonic Bone Scalpel Group | Standard of Care Group
Number analyzed (Participants) | 30 | 30
grams/deciliter | 30.39 (10.7) | 30.45 (9.51)

12. Other Pre Specified Outcome: Intraoperative Use of Antifibrinolytic
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasonic Bone Scalpel Group | Standard of Care Group
Number analyzed (Participants) | 32 | 33
Participants | 32 | 33

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Ultrasonic Bone Scalpel Group | Standard of Care Group
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT02781324/Prot_SAP_000.pdf